CLINICAL TRIAL: NCT00477308
Title: Clinical, Immunologic and Virological Outcomes of Genotyping Directed Salvage Therapy in Children Who Have Failed Dual NRTIs
Brief Title: Genotyping Directed Salvage Therapy in Children Who Have Failed Dual NRTIs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Swiss Cohort (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 013 phase II
Record Dates: First submitted 2007-05-20; First posted 2007-05-23 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: HIV children; genotypic resistance; dual NRTIs; Salvage therapy; treatment outcome; Salvage therapy based on genotyping results; Treatment Failure
MeSH Terms: conditions — HIV Infections | interventions — Salvage Therapy

STUDY DESIGN:
Intervention Model Description: salvage therapy
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- salvage therapy (Other): Children with drug resistance were treated using the drug resistant profile
  Interventions: Procedure: salvage therapy

INTERVENTIONS:
Procedure: salvage therapy

SUMMARY:
In HIV-NAT 013 phase I study, genotyping was performed in 95 children on dual NRTI which showed that almost all children had resistance to NRTi. The HIV-NAT 013 phase II is a follow up study to evaluate treatment outcome after salvage therapy and the evolution of mutations.

DETAILED DESCRIPTION:
The HIV-NAT 013 study (conducted in 2003) evaluated prevalence and pattern of RT mutation in 95 children treated with dual NRTI. The study showed almost all children to have some degree of NRTI resistance and 40% with multi NRTI resistance. The mutation reported was major mutation.

After the study, the patients were managed based on the physician's judgment using genotyping results. The 95 patients in HIV-NAT 013 are categorized into 3 groups.

1. No viral resistance
2. Low grade resistance with or without clinical/ immunological failure
3. High grade resistance with or without clinical/ immunological failure.

There are limited prospective studies evaluating outcome of decision regarding salvage therapy after genotyping results

There are also new mutations that are not considered major mutation that may affect treatment outcome

Knowledge learned from this study will benefit Thai children with NRTI resistance by helping pediatricians better choose salvage treatment options

ELIGIBILITY:
Inclusion Criteria:

* All children from HIV-NAT 013 phase I

Exclusion Criteria:

* No inform consent obtained

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2006-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Clinical, immunologic and virologic outcome of children who had genotyping directed salvage therapy | 1 time point (Cross Sectional Study)

SECONDARY OUTCOMES:
Comparison outcome of children in the 3 groups, | 1 time point
Changes of mutation in children within the 3 groups, and | 1 time point
Effect of previously unreported mutations, minor and others, on treatment outcome | 1 time point

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT); Tawee Chotpitayasunondh, MD, Principal Investigator — Queen Sirikit National Institute of Child Health, Bangkok
Locations (3):
- Thailand (3):
  - Chulalongkorn Hospital, Bangkok
  - Queen Sirikit National Institute of Child Health, Bangkok, Bangkok
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok

REFERENCES:
- [Result] Bunupuradah T, Suntarattiwong P, Li A, Sirivichayakul S, Pancharoen C, Boonrak P, Puthanakit T, Kerr SJ, Ruxrungtham K, Chotpitayasunondh T, Hirschel B, Ananworanich J; HIV-NAT 013 Study Team. Antiretroviral treatment outcome following genotyping in Thai children who failed dual nucleoside reverse transcriptase inhibitors. Int J Infect Dis. 2010 Apr;14(4):e311-6. doi: 10.1016/j.ijid.2009.05.017. Epub 2009 Aug 21. PMID 19699673
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org